CLINICAL TRIAL: NCT07297446
Title: Phenotypic and Functional Profile of Peripheral Blood Lymphomonocytes in Seborrheic Dermatitis.
Acronym: PHENOTYPIC
Status: Completed | Type: Observational
Sponsor: San Gallicano Dermatological Institute IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: RS 170/ISG/24
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Seborrheic Dermatitis; Dietary Habits
Keywords: phenotypic and functional profile; peripheral-blood lymphomonocytes; seborrheic dermatitis (SD)
MeSH Terms: conditions — Dermatitis, Seborrheic; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Seborrheic Dermatitis (DS): Participants aged 45-75 years with mild-to-moderate facial seborrheic dermatitis. Additional sebaceous areas may be affected. Blood samples are collected for plasma analysis (secretory and lipidomic profiling) and for lymphomonocyte isolation and flow cytometric phenotyping. Participants also complete a dietary habits questionnaire.
- Non-Affected Controls (NA): Healthy volunteers aged 45-75 years with no seborrheic dermatitis or other relevant dermatologic diseases. Controls undergo the same laboratory and questionnaire procedures as the DS group.

SUMMARY:
The protocol describes a prospective, monocentric pilot study conducted at the Istituto Dermatologico San Gallicano (IFO-ISG) aimed at investigating the phenotypic and functional profile of peripheral-blood lymphomonocytes in individuals with seborrheic dermatitis (SD) compared with non-affected controls. A secondary objective is to explore dietary habits in subjects with SD.

Seborrheic dermatitis is a chronic-relapsing inflammatory skin disease, common in infancy, puberty, and adulthood (40-60 years). Its multifactorial etiology involves:

Sebaceous gland hyperactivity and altered lipid composition promoting Malassezia proliferation;

Metabolic activation of sebaceous glands by Malassezia, which generates irritating fatty acids;

Immune dysregulation, influencing keratinocyte activation and differentiation;

Barrier disruption, clinically resulting in erythema, scaling, and pruritus.

Previous research on immune cells in barrier tissues (gut, lung, skin) suggests that environmental factors-particularly dietary fatty acids and salt intake-modulate the functional polarization of Th17 vs. Treg cells, with implications for autoimmunity. Tissue-resident memory T cells (TRM), abundant in barrier organs, display site-specific homing markers such as CCR4, CCR10, CXCR4, GATA6, and BCL6. In contrast, circulating TEM and TEMRA subsets share common profiles across tissues.

Protocollo_Profilo fenotipico e…

In skin, Th17 cells exhibit variable transcriptional states that may reflect tissue-dependent functional states rather than fixed subtypes. Studies in SD have mainly focused on cutaneous immune responses, highlighting roles for Tγδ cells, cytokines (IL-1α, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-17, TNF-α), and β-defensins, linked to dendritic-cell maturation driven by sebaceous lipids and activation of the NLRP3 inflammasome. Malassezia can also induce IL-1β release from dendritic cells in vitro. However, little is known about how SD affects circulating immune cells or how dietary patterns influence systemic immune responses in this disease.

Study population

The study will include 15 SD patients and 15 non-affected (NA) controls, aged 45-75 years, of both sexes. SD patients must have mild-to-moderate facial involvement and must have stopped topical or systemic treatments for at least two weeks. Exclusion criteria include other skin diseases, neurodegenerative disorders, immunosuppression, ongoing treatments, or HIV positivity. Controls are selected from IFO staff, relatives, and individuals undergoing routine dermatologic examinations.

Methods

After overnight fasting, participants undergo venous blood sampling (7 mL). Plasma is separated and stored at -80°C for secretory and lipidomic profiling. Lymphomonocytes are isolated using Ficoll-Hypaque gradients and analyzed by flow cytometry to characterize immunological phenotypes. Each participant completes a dietary questionnaire at enrollment. Collected data include demographics, clinical history, dietary information, laboratory findings, and SD-specific clinical data (for the patient group).

Statistical plan

As a pilot study, data will be summarized with descriptive statistics only; no formal comparisons will be performed. Findings will generate hypotheses for future research. Recruitment is planned over 18 months, with a total study duration of 24 months.

Ethical and administrative aspects

The study adheres to Good Clinical Practice, the Declaration of Helsinki, and EU/national regulations. Ethical approval is required before initiation. Participants must provide written informed consent for both study participation and data processing. Data will be handled in compliance with GDPR, using pseudonymization, secure storage, and restricted access. Authorized monitors and regulatory authorities may inspect source documents. Biologic samples will be stored until completion of analyses. Results will be published in aggregated, non-identifiable form in scientific journals and conferences.

DETAILED DESCRIPTION:
Seborrheic dermatitis (SD) is a chronic-relapsing inflammatory skin disease with three incidence peaks: within the first three months of life, during puberty, and in adulthood (40-60 years). Its etiology is multifactorial and can be attributed to: (I) excessive sebum production by the sebaceous gland (SG) and alterations in its composition, creating an environment favorable to the growth of Malassezia; (II) activation of SG metabolism and its secretory activity by Malassezia, with the release of irritating saturated and unsaturated fatty acids; (III) impaired immune system function, leading to the induction of keratinocyte activation and differentiation; and (IV) disruption of the skin barrier, responsible for clinical manifestations such as erythema, itching, and scaling.

Studies focusing on the presence of immunocompetent cells at barrier sites (intestinal lamina propria, lungs, and skin) have shown that, at the intestinal level, diet and metabolism can influence the phenotype of Th17 lymphocytes. Indeed, dietary enrichment in short-chain fatty acids can promote differentiation toward Treg, whereas the habitual dietary intake of long-chain fatty acids, as well as higher salt consumption, is associated with an increased number of lymphocytes with a Th17 functional profile, and thus with a state of autoimmunity. Barrier sites are typically rich in TRM (tissue-resident memory T) cells, which display site-specific functional profiles tailored to local homing requirements. In the skin, TRM are characterized by high expression of CCR4, CCR10, CXCR4, GATA6, and BCL6. In contrast, the TEM (T effector memory) and TEMRA (terminally differentiated effector memory) compartments appear to share a functional profile across different barrier sites and peripheral tissues.

However, the classification of barrier-site T cells into Th1, Th17, and Th2 subtypes should be viewed in a nuanced way-as an expression of functional characteristics rather than the final outcome of a maturation and differentiation process. In particular, Th17 lymphocytes can modify their functional phenotype, exhibiting distinct transcriptional profiles associated with either homeostatic or pathogenic potential, suggesting that these should be considered tissue-dependent functional states rather than different cell types. Th17 lymphocytes are associated with secretion of IL-17A, IL-17F, and IL-22, and depend on the RORγt-dependent signaling pathway, while TGF-β and IL-6 are required for their generation from naïve T lymphocytes. Studies on the involvement of immune components in the etiopathogenesis of SD have so far focused on the skin, where a role for γδ T cells has been observed, with secretion of IL-1α, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-17, TNF-α, β-defensins-likely related to the maturation of dendritic cells induced by sebaceous lipids and the subsequent induction of the NLRP3 inflammasome.

Malassezia itself can induce the release of IL-1β in vitro by dendritic cells obtained from peripheral blood.

No studies are currently available on the possible involvement, in terms of functional modulation, of peripheral blood lymphomonocytes in the pathogenesis of SD.

Likewise, despite known dietary influences on Th17 cell function at barrier sites such as the intestinal mucosa, data are lacking regarding the role of diet and lifestyle in seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Facial Seborrheic Dermatitis (SD) of mild to moderate severity; other sebaceous areas of the body may also be affected.

Both sexes. Age 45-75 years. Treatments for SD, topical and/or systemic, suspended for at least two (2) weeks.

Willingness to comply with the appointments/procedures required by the study. Signature of the informed consent.

Exclusion Criteria:

* Concomitant dermatological conditions, such as, for example, atopic dermatitis, rosacea, acne, psoriasis, besides the inclusion condition (Seborrheic Dermatitis).

Diagnosed neurodegenerative diseases. Ongoing pharmacological treatment, topical or systemic, for Seborrheic Dermatitis (SD).

Immunosuppression. HIV seropositivity.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of people affected by SD (Seborrheic Dermatitis), both female and male, aged between 45 and 75 years, and healthy subjects selected from personnel undergoing routine examinations by the IFO Occupational Health Unit (Medicina del Lavoro IFO) and among members, friends, and relatives of the personnel of the Cutaneous Physiopathology Unit (UOC Fisiopatologia Cutanea).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Phenotypic and Functional Profile of Peripheral Blood Lymphomonocytes | Baseline (Day 1)
  Evaluation of the immunological profile of Peripheral Blood Mononuclear Cells (PBMCs) in patients with Seborrheic Dermatitis compared to healthy controls. The analysis includes:
  Phenotypic Characterization (Flow Cytometry): Expression of cell surface markers to identify Regulatory T cells (CD45, CD4, CD25, CD127, FoxP3), general immune subsets (CD3, CD4, CD8, CD14, CD16, CD19, CD45, CD56), and activated T cells (CD8, HLA-DR, CD38, CD3, CD4, CD45RA, CD197).
  Functional/Secretory Profile (Multiplex/ELISA): Measurement of plasma concentrations of the following cytokines: IL-4, IL-5, IL-8, IL-12, IL-13, IL-18, IL-31, TNF-a, IFN-a, IFN-g, GRO-a, IL-6, IL1a/b, IL-20, IL-23, IL-17A/F, IL-22, GM-CSF, and TSLP.

SECONDARY OUTCOMES:
Assessment of Dietary Habits | Baseline (Day 1)
  Evaluation of dietary habits and lifestyle through a self-administered food frequency and lifestyle questionnaire (including elements of the MeDiWeB questionnaire) to compare nutritional patterns between the Seborrheic Dermatitis group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- San Gallicano Dermatological Institute IRCCS, Roma, Italy, Italy